CLINICAL TRIAL: NCT04782128
Title: A Randomized, Open-label, Multicenter Study of the Efficacy and Safety of RC28-E Injection in Subjects With Moderately Severe to Severe Nonproliferative Diabetic Retinopathy
Brief Title: Evaluation of RC28-E Injection in Diabetic Retinopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 28C003
Record Dates: First submitted 2021-03-01; First posted 2021-03-04 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — RC28-E protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- intravitreal 1.0mg RC28-E injection Q8 (Experimental): Subjects received 1.0mg intravitreal RC28-E injection every 4 weeks for 3 visits followed by injections every 8 weeks.
  Interventions: Biological: RC28-E injection
- Experimental: intravitreal 1.0mg RC28-E injection PRN (Experimental): Subjects received 1.0mg intravitreal RC28-E injection every 4 weeks for 5 visits followed by injections an as needed (PRN) schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: RC28-E injection
- Experimental: intravitreal 2.0mg RC28-E injection Q8 (Experimental): Subjects received 2.0mg intravitreal RC28-E injection every 4 weeks for 3 visits followed by injections every 8 weeks.
  Interventions: Biological: RC28-E injection
- Experimental: intravitreal 2.0mg RC28-E injection PRN (Experimental): Subjects received 1.0mg intravitreal RC28-E injection every 4 weeks for 5 visits followed by injections an as needed (PRN) schedule based upon the physician assessment in accordance with pre-specified criteria.
  Interventions: Biological: RC28-E injection

INTERVENTIONS:
Biological: RC28-E injection — a chimric decoy receptor trap fusion protein by dual blockage of VEGF and FGF

SUMMARY:
This is a randomized, open-label, multicenter study of the efficacy and safety of RC28-E injection (a chimric decoy receptor trap fusion protein by dual blockage of VEGF and FGF-2) in the treatment of patients with moderately severe to severe nonproliferative diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Sign the consent form, willing and able to comply with clinic visits and study-related procedures;
* Aged 18 years to 80 years, male or female;
* Diabetes mellitus(type 1 or 2);
* Moderately severe to severe NPDR (DRSS levels 47 or 53) which was confirmed by the central reading center, and in whom PRP can be safely deferred by the investigator's judgement;
* BCVA score in the study eye of ≥69 letters (approximate Snellen equivalent of 20/40 or better) using the ETDRS protocol at an initial testing distance of 4 meters;
* If both eyes meet the inclusion criterion, one eye with poor BCVA is selected as the study eye;

Exclusion Criteria:

* Presence of DME threatening the center of the macula (within 1,000 microns of the foveal center) in the study eye;
* Evidence of retinal neovascularization on clinical examination or FA;
* Any prior focal or grid laser photocoagulation (within 1,000 microns of the foveal center) or PRP in the study eye;
* Current ASNV, vitreous hemorrhage, tractional retinal detachment or epiretinal membrane involved the macular in the study eye;
* History of vitreoretinal surgery in the study eye;
* Active infectious blepharitis, keratitis, scleritis, conjunctivitis at the screening assessments in either eye ;
* Previous treatment with anti-angiogenic drugs in either eye or system (ranibizumab, aflibercept, conbercept, etc) within 3 months of the Day 0 visit;
* Previous use of intraocular or periocular corticosteroids (such as triamcinolone acetonide, dexamethasone vitreous implant) in either eye within 6 months of day 0.
* Uncontrolled clinical disease (such as severe psychiatric, neurological, cardiovascular, respiratory disease or other systemic diseases) and tumors;
* Pregnant or lactating women, subjects who had family planning throughout the study period;
* Those who participated in clinical trials for 3 months or 5 half-lives of the investigational product (the longer the time) before theDay 0
* Those who considered unsuitable for enrollment by investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who have improved by ≥2 steps from baseline in DRSS score at week 24, 52 | At Week 24, 52
  The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at week 24, 52 from baseline

SECONDARY OUTCOMES:
Percentage of Participants Who Developed a Vision-Threatening Complication Due to Diabetic Retinopathy at Week 24, 52 | At Week 24, 52
  Vision-threatening complications are defined as the composite outcome of proliferative diabetic retinopathy (inclusive of participants who have vitreous hemorrhage or tractional retinal detachment believed to be due to PDR) and anterior segment neovascularization (ASNV) (participants with neovascularization of the iris and/or definitive neovascularization of the iridocorneal angle).
Percentage of Participants Who Developed Central Involved-Diabetic Macular Edema (CI-DME) at Week 24, 52; | At Week 24, 52
  The percentage of participants who developed CI-DME at week24, 52 were reported.
Mean Change from Baseline in Best Corrected Visual Acuity (BCVA); | Baseline up to week 52
  Measurement of visual acuity with Early Treatment Diabetic Retinopathy Study (ETDRS) charts.
Mean change from baseline in DRSS score; | Baseline upto week 52
  The Diabetic Retinopathy Disease Severity Scale (DRSS) may be used to describe overall retinopathy severity as well as the change in severity over time. Here, DRSS describes severity level 47 (moderately severe NPDR) and level 53 (severe NPDR) at week 24, 52 from baseline.
Percentage of Participants Who Received Panretinal Photocoagulation (PRP) at Week24, 52; | At Week 24, 52
  The percentage of participants who received panretinal photocoagulation (PRP).
Percentage of participants who undergoing Vitrectomy at Week24, 52; | At Week 24, 52
  The percentage of participants who undergoing vitrectomy.
Frequency of administration RC28-E; | At Week 24, 52
  Number of intravitreal injections
Safety of RC28-E injection | Baseline upto week 52
  Incidence of AE in ocular and non-ocular

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided